CLINICAL TRIAL: NCT00624780
Title: Long Term Safety And Efficacy Study Of Pregabalin (Lyrica) In Subjects With Generalized Anxiety Disorder
Brief Title: Safety and Efficacy Evaluation Of Pregabalin (Lyrica) With Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081147
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2012-09

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Pregabalin; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Pregabalin
- 2 (Active Comparator)
  Interventions: Drug: Lorazepam
- 3 (Experimental)
  Interventions: Drug: Pregabalin
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150-300 mg given twice a day
  Other Names: Lyrica
  Arms: 1
Drug: Lorazepam — Lorazepam 3-4 mg given twice a day
  Arms: 2
Drug: Pregabalin — Pregabalin 450-600 mg given twice a day
  Other Names: Lyrica
  Arms: 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
The purpose of this study is to characterize the safety and efficacy in patients with generalized anxiety disorder after short- (3 months) and long-term (6 months) use of Pregabalin (Lyrica).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Generalized Anxiety Disorder
* HAM-A score >=18 and HAM-D (item 1) score >=2 at screening and baseline
* Needs pharmacological treatment

Exclusion Criteria:

* Current or past diagnosis of any other DSM IV Axis I disorders
* A history of failed treatment with a benzodiazepine
* Any clinically significant, serious, or unstable hematologic, autoimmune, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- Argentina (3):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Lanús, Prov. de Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Pfizer Investigational Site, Vienna, Austria
- Pfizer Investigational Site, San José, Costa Rica
- Croatia (3):
  - Pfizer Investigational Site, Rijeka
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Zagreb
- Czechia (8):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Litoměřice
  - Pfizer Investigational Site, Lnáře
  - Pfizer Investigational Site, Mělník
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 10- Strasnice
  - Pfizer Investigational Site, Strakonice
- Finland (6):
  - Pfizer Investigational Site, Espoo
  - Pfizer Investigational Site, HUS
  - Pfizer Investigational Site, Joensuu
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Seinäjoki
  - Pfizer Investigational Site, Turku
- Pfizer Investigational Site, Athens, Greece
- India (5):
  - Pfizer Investigational Site, Ellisbridge, Ahmedabad
  - Pfizer Investigational Site, Tirupati, Andhra Pradesh
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Indonesia (4):
  - Pfizer Investigational Site, Denpasar, Bali
  - Pfizer Investigational Site, Jakarta, Jakarta Selatan
  - Pfizer Investigational Site, Jakarta Selatan, Jakarta Special Capital Region
  - Pfizer Investigational Site, Surabaya
- Lithuania (3):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Klaipėda
  - Pfizer Investigational Site, Vilnius
- Mexico (3):
  - Pfizer Investigational Site, Acapulco de Juárez, Guerrero
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Mexico City
- Russia (3):
  - Pfizer Investigational Site, Khotkovo, Moscow Region
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Kragujevac
- Pfizer Investigational Site, Ljubljana, Slovenia
- Spain (2):
  - Pfizer Investigational Site, Langreo, Principality of Asturias
  - Pfizer Investigational Site, Zamora
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Kocaeli

REFERENCES:
- [Derived] Kasper S, Iglesias-Garcia C, Schweizer E, Wilson J, DuBrava S, Prieto R, Pitman VW, Knapp L. Pregabalin long-term treatment and assessment of discontinuation in patients with generalized anxiety disorder. Int J Neuropsychopharmacol. 2014 May;17(5):685-95. doi: 10.1017/S1461145713001557. Epub 2013 Dec 19. PMID 24351233

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study employed 3 treatments in Period 1 and 6 treatments in Period 2. Randomization occurred once, at the onset of Period 1.
Groups:
- Pregabalin High Dose, Pregabalin High Dose: Period 1 (treatment optimization): Pregabalin capsule 150 milligram per day (mg/day) orally twice daily in 2 equally divided doses in Week 1, pregabalin capsule 300 mg/day orally twice daily in 2 equally divided doses in Week 2 and pregabalin capsule 450 mg/day orally twice daily in 2 equally divided doses in Week 3 during 3-week upward titration. Flexible dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses up to Week 12. Period 2 (fixed dosing): Continued pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses up to Week 24. Period 3 (treatment discontinuation): A 1-week blinded dose tapering period (Week 25). Participants were followed-up after 1 week (Week 26).
- Pregabalin High Dose, Placebo: Period 1 (treatment optimization): Pregabalin capsule 150 mg/day orally twice daily in 2 equally divided doses in Week 1, pregabalin capsule 300 mg/day orally twice daily in 2 equally divided doses in Week 2 and pregabalin capsule 450 mg/day orally twice daily in 2 equally divided doses in Week 3 during 3-week upward titration. Flexible dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses up to Week 12. Period 2 (fixed dosing): Pregabalin was discontinued with a blinded dose tapering over 1-week followed by matching placebo capsule orally twice daily up to Week 24. Period 3 (treatment discontinuation): Continued matching placebo capsule orally twice daily for 1 week (Week 25). Participants were followed-up after 1 week (Week 26).
- Pregabalin Low Dose, Pregabalin Low Dose: Period 1 (treatment optimization): Pregabalin capsule 150 mg/day orally twice daily in 2 equally divided doses during 3-week upward titration. Flexible dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses up to Week 12. Period 2 (fixed dosing): Continued pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses up to Week 24. Period 3 (treatment discontinuation): A 1-week blinded dose tapering period (Week 25). Participants were followed-up after 1 week (Week 26).
- Pregabalin Low Dose, Placebo: Period 1 (treatment optimization): Pregabalin capsule 150 mg/day orally twice daily in 2 equally divided doses during 3-week upward titration. Flexible dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses up to Week 12. Period 2 (fixed dosing): Pregabalin was discontinued with a blinded dose tapering over 1-week followed by matching placebo capsule orally twice daily up to Week 24. Period 3 (treatment discontinuation): Continued matching placebo capsule orally twice daily for 1 week (Week 25). Participants were followed-up after 1 week (Week 26).
- Lorazepam, Lorazepam: Period 1 (treatment optimization): Lorazepam capsule 2 mg/day orally twice daily in 2 equally divided doses in Week 1, lorazepam capsule 3 mg/day orally in 2 divided doses (1 mg in morning, 2 mg at night) in Week 2 and 3, during 3-week upward titration. Flexible dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) up to Week 12. Period 2 (fixed dosing): Continued lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) up to Week 24. Period 3 (treatment discontinuation): A 1-week blinded dose tapering period (Week 25). Participants were followed-up after 1 week (Week 26).
- Lorazepam, Placebo: Period 1 (treatment optimization): Lorazepam capsule 2 mg/day orally twice daily in 2 equally divided doses in Week 1, lorazepam capsule 3 mg/day orally in 2 divided doses (1 mg in morning, 2 mg at night) in Week 2 and 3, during 3-week upward titration. Flexible dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) up to Week 12. Period 2 (fixed dosing): Lorazepam was discontinued with a blinded dose tapering over 1-week followed by matching placebo capsule orally twice daily up to Week 24. Period 3 (treatment discontinuation): Continued matching placebo capsule orally twice daily for 1 week (Week 25). Participants were followed-up after 1 week (Week 26).
Period: Treatment Optimization (Up to Week 12)
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Started | 154 | 52 | 154 | 52 | 153 | 50
Completed | 121 | 39 | 112 | 38 | 114 | 39
Not Completed | 33 | 13 | 42 | 14 | 39 | 11
Not completed — Adverse Event | 7 | 5 | 15 | 3 | 9 | 5
Not completed — Lack of Efficacy | 5 | 2 | 10 | 5 | 9 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 10 | 2 | 7 | 4 | 10 | 4
Not completed — Other | 10 | 4 | 8 | 2 | 9 | 0
Period: Fixed Dosing (Week 13 to Week 24)
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Started | 121 | 39 | 112 | 38 | 114 | 39
Completed | 106 | 28 | 94 | 27 | 95 | 30
Not Completed | 15 | 11 | 18 | 11 | 19 | 9
Not completed — Adverse Event | 5 | 4 | 5 | 2 | 3 | 1
Not completed — Lack of Efficacy | 2 | 1 | 2 | 5 | 5 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 6 | 3 | 6 | 2
Not completed — Other | 5 | 3 | 4 | 1 | 4 | 3
Period: Treatment Discontinuation (Week 25)
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Started | 106 | 28 | 94 | 27 | 95 | 30
Completed | 104 | 28 | 91 | 26 | 95 | 29
Not Completed | 2 | 0 | 3 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Period: Follow-up (Week 26)
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Started | 104 | 28 | 91 | 26 | 95 | 29
Completed | 102 | 27 | 89 | 26 | 93 | 29
Not Completed | 2 | 1 | 2 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo | Total
Number analyzed (Participants) | 154 | 52 | 154 | 52 | 153 | 50 | 615
Age, Customized [Number; unit: participants]
  18 to 44 years | 75 | 30 | 100 | 28 | 86 | 27 | 346
  45 to 64 years | 79 | 22 | 51 | 24 | 66 | 23 | 265
  Greater than or equal to 65 years | 0 | 0 | 3 | 0 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 30 | 101 | 32 | 95 | 27 | 374
  Male | 65 | 22 | 53 | 20 | 58 | 23 | 241

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 1
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms; 14 item questionnaire scored 0 (not present) to 4 (very severe); total possible range 0 to 56. Lower score indicates less affected.
Time Frame: Baseline, Week 1 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included. n=participants evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pregabalin High Dose: Period 1 (treatment optimization): Pregabalin capsule 150 milligram per day (mg/day) orally twice daily in 2 equally divided doses in Week 1, pregabalin capsule 300 mg/day orally twice daily in 2 equally divided doses in Week 2 and pregabalin capsule 450 mg/day orally twice daily in 2 equally divided doses in Week 3 during 3-week upward titration. Flexible dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 450 mg/day or 600 mg/day orally twice daily in 2 equally divided doses up to Week 12.
- Pregabalin Low Dose: Period 1 (treatment optimization): Pregabalin capsule 150 mg/day orally twice daily in 2 equally divided doses during 3-week upward titration. Flexible dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses up to Week 12.
- Lorazepam: Period 1 (treatment optimization): Lorazepam capsule 2 mg/day orally twice daily in 2 equally divided doses in Week 1, lorazepam capsule 3 mg/day orally in 2 divided doses (1 mg in morning, 2 mg at night) in Week 2 and 3, during 3-week upward titration. Flexible dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6, fixed dosing of lorazepam capsule 3 or 4 mg/day orally twice daily in 2 divided doses (1 or 2 mg in morning, 2 mg at night) up to Week 12.
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 19 | 21
units on a scale
  Baseline (n=15,19,21) | 25.8 (4.23) | 24.9 (4.15) | 24.4 (4.88)
  Change at Discontinuation Week 1 (n=15,19,18) | -7.7 (6.75) | -5.9 (7.20) | -9.9 (10.81)

2. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 2
Description: as for outcome 1
Time Frame: Baseline, Week 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included in less-than Month 3 last visit analysis. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 14 | 15 | 16
units on a scale | -12.0 (7.24) | -5.9 (5.46) | -9.7 (11.08)

3. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 2 (3-Month Last Visit) at Discontinuation Week 1
Description: as for outcome 1
Time Frame: Baseline, Week 1 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. Cohort 2: Participants who discontinued study from Week 9 to Week 15 and had at least 1 discontinuation assessment were included in Month 3 last visit analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 52
units on a scale
  Baseline | 25.0 (5.37) | 24.7 (3.89) | 24.6 (4.76)
  Change at Discontinuation Week 1 | -15.3 (7.76) | -15.3 (6.71) | -15.8 (7.92)

4. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 2 (3-Month Last Visit) at Discontinuation Week 2
Description: as for outcome 1
Time Frame: Baseline, Week 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: Per-protocol analysis set. Cohort 2: Participants who discontinued study from Week 9 to Week 15 and had at least 1 discontinuation assessment were included in Month 3 last visit analysis. Here, N (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 54 | 49 | 44
units on a scale | -15.6 (7.42) | -14.9 (7.11) | -16.0 (7.96)

5. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 3 (6-Month Last Visit) at Discontinuation Week 1
Description: as for outcome 1
Time Frame: Baseline, Week 1 post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included in Month 6 last visit analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pregabalin Low Dose, Placebo: Period 1 (treatment optimization): Pregabalin capsule 150 mg/day orally twice daily in 2 equally divided doses during 3-week upward titration. Flexible dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses depending on efficacy and tolerability up to Week 6. If participant had an adequate response at Week 6 fixed dosing of pregabalin capsule 150 mg/day or 300 mg/day orally twice daily in 2 equally divided doses up to Week 12. Period 2 (fixed dosing): Pregabalin was discontinued with a blinded dose tapering over 1-week followed by matching placebo capsule orally twice daily up to Week 24. Period 3 (treatment discontinuation): Continued matching placebo capsule orally twice daily for 1 week (Week 25). Participants were followed-up after 1 week (Week 26).
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 29 | 100 | 30
units on a scale
  Baseline | 25.5 (3.85) | 24.2 (4.64) | 24.7 (3.85) | 24.9 (3.82) | 24.6 (4.36) | 24.9 (3.93)
  Change at Discontinuation Week 1 | -17.6 (7.25) | -18.7 (5.36) | -18.4 (6.33) | -16.5 (7.25) | -16.2 (8.11) | -19.1 (6.69)

6. Primary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) for Cohort 3 (6-Month Last Visit) at Discontinuation Week 2
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms; 14 item questionnaire scored 0 (not present) to 4 (very severe); possible range 0 to 56. Lower score indicates less affected.
Time Frame: Baseline, Week 2 post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included in Month 6 last visit analysis. Here, N (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 107 | 29 | 84 | 26 | 94 | 30
units on a scale | -16.6 (8.53) | -19.1 (5.80) | -18.3 (7.05) | -16.0 (8.17) | -16.7 (7.52) | -18.7 (7.38)

7. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 1
Description: PWC: 20 item physician rated interview measuring anxiolytic drug withdrawal-related signs and symptoms (gastrointestinal, mood, sleep, motor, somatic, perception and cognition); range 0 (not present) to 3 (severe); total score range: 0 to 60; higher score = more affected.
Time Frame: Last visit on treatment, Week 1 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included in less-than Month 3 last visit analysis. N (Number of Participants Analyzed) = participants evaluable for this measure. 'n' = participants evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 18 | 20
units on a scale
  Last visit on treatment (n=15,18,20) | 10.1 (8.72) | 16.8 (13.20) | 13.1 (10.75)
  Change at Discontinuation Week 1 (n=15,18,18) | 0.1 (9.89) | -2.8 (7.99) | -4.2 (6.12)

8. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 2
Description: as for outcome 7
Time Frame: Last visit on treatment, Week 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included in less-than Month 3 last visit analysis. Here, N (Number of Participants Analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 14 | 15 | 16
units on a scale | -2.0 (6.39) | -2.7 (9.04) | -3.2 (6.05)

9. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 2 (3-Month Last Visit) at Discontinuation Week 1
Description: as for outcome 7
Time Frame: Last visit on treatment, Week 1 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 50
units on a scale
  Last visit on treatment | 7.2 (7.32) | 6.5 (6.01) | 5.0 (3.80)
  Change at Discontinuation Week 1 | 1.9 (7.29) | 1.4 (4.52) | 2.3 (6.60)

10. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 2 (3-Month Last Visit) at Discontinuation Week 2
Description: as for outcome 7
Time Frame: Last visit on treatment, Week 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 54 | 49 | 44
units on a scale | 2.1 (6.11) | 2.0 (5.51) | 1.6 (6.33)

11. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 3 (6-Month Last Visit) at Discontinuation Week 1
Description: as for outcome 7
Time Frame: Last visit on treatment, Week 1 post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included in Month 6 last visit analysis. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 93 | 29 | 100 | 30
units on a scale
  Last visit on treatment | 5.2 (5.62) | 4.9 (7.15) | 3.9 (4.14) | 6.5 (6.72) | 5.3 (6.65) | 4.7 (4.50)
  Change at Discontinuation Week 1 | 1.7 (4.92) | 0.0 (2.18) | 1.1 (3.50) | 1.0 (4.37) | 3.0 (6.79) | -0.1 (3.22)

12. Primary Outcome: Change From Last Visit on Treatment in Physician's Withdrawal Checklist (PWC) Score for Cohort 3 (6-Month Last Visit) at Discontinuation Week 2
Description: as for outcome 7
Time Frame: Last visit on treatment, Week 2 post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 106 | 29 | 84 | 26 | 93 | 30
units on a scale | 2.8 (5.99) | -1.0 (5.65) | 1.7 (4.78) | 1.8 (5.14) | 2.2 (6.02) | -0.1 (3.63)

13. Secondary Outcome: Number of Participants With Rebound Anxiety for Cohort 1 (Less Than 3-Month Last Visit)
Description: Rebound anxiety was defined as a rapid return of the participant's original symptoms following drug discontinuation, that were worse compared to baseline. This was characterized by a HAM-A score at the Discontinuation Week 1 or Week 2 greater than or equal to the baseline value.
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included in less-than Month 3 last visit analysis. Here, N (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 19 | 18
participants | 1 | 5 | 1

14. Secondary Outcome: Number of Participants With Rebound Anxiety for Cohort 2 (3-Month Last Visit)
Description: as for outcome 13
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 48
participants | 3 | 1 | 2

15. Secondary Outcome: Number of Participants With Rebound Anxiety for Cohort 3 (6-Month Last Visit)
Description: as for outcome 13
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 28 | 100 | 30
participants | 4 | 0 | 0 | 1 | 6 | 0

16. Secondary Outcome: Number of Participants With Discontinuation-Emergent Signs and Symptoms (DESS) for Cohort 1 (Less Than 3-Month Last Visit)
Description: DESS adverse events, a subset of Treatment Emergent Signs and Symptoms (TESS), were defined as those spontaneously reported adverse events that developed or existed prior to but worsened during Discontinuation Week 1 and 2.
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study prior to Week 9 and had at least 1 discontinuation assessment were included in less-than Month 3 last visit analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 19 | 21
participants
  Newly developed DESS | 6 | 0 | 3
  Worsened DESS | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Discontinuation-Emergent Signs and Symptoms (DESS) for Cohort 2 (3-Month Last Visit)
Description: as for outcome 16
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: Per-protocol analysis set. Cohort 1: Participants who discontinued study from Week 9 to Week 15 and had at least 1 discontinuation assessment were included in Month 3 last visit analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 52
participants
  Newly developed DESS | 40 | 38 | 36
  Worsened DESS | 1 | 2 | 1

18. Secondary Outcome: Number of Participants With Discontinuation-Emergent Signs and Symptoms (DESS) for Cohort 3 (6-Month Last Visit)
Description: as for outcome 16
Time Frame: 2 weeks post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included in Month 6 last visit analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 29 | 100 | 30
participants
  Newly developed DESS | 78 | 5 | 35 | 17 | 50 | 7
  Worsened DESS | 2 | 0 | 2 | 1 | 5 | 0

19. Secondary Outcome: Change From Baseline in Physician's Withdrawal Checklist (PWC) Score for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 7
Time Frame: Baseline, Week 1, 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 14 | 19 | 21
units on a scale
  Baseline (n=14,19,21) | 13.6 (8.19) | 17.6 (10.68) | 16.4 (8.62)
  Change at Discontinuation Week 1 (n=14,19,18) | -3.4 (11.91) | -3.3 (9.12) | -5.9 (7.43)
  Change at Discontinuation Week 2 (n=13,15,16) | -4.7 (10.62) | -2.7 (8.20) | -5.4 (8.34)

20. Secondary Outcome: Change From Baseline in Physician's Withdrawal Checklist (PWC) Score for Cohort 2 (3-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 7
Time Frame: Baseline, Week 1, 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: Per-protocol analysis set. Cohort 2: Participants who discontinued study from Week 9 to Week 15 and had at least 1 discontinuation assessment were included in Month 3 last visit analysis. N (Number of Participants Analyzed) = participants evaluable for this measure. 'n' = participants evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 57 | 51 | 52
units on a scale
  Baseline (n=57,51,52) | 17.4 (7.81) | 17.1 (9.84) | 14.8 (7.86)
  Change at Discontinuation Week 1 (n=57,51,49) | -8.5 (9.40) | -9.3 (9.48) | -7.6 (9.53)
  Change at Discontinuation Week 2 (n=53,48,44) | -8.3 (9.53) | -8.7 (9.68) | -8.0 (9.70)

21. Secondary Outcome: Change From Baseline in Physician's Withdrawal Checklist (PWC) Score for Cohort 3 (6-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 7
Time Frame: Baseline, Week 1, 2 post-treatment discontinuation (discontinuation [DC] occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included. N (Number of Participants Analyzed) = participants evaluable for this measure. 'n'=participants evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 29 | 99 | 30
units on a scale
  Baseline (n=109,30,94,29,99,30) | 17.8 (8.36) | 17.8 (7.79) | 16.1 (7.52) | 17.4 (9.28) | 16.8 (8.85) | 14.9 (7.61)
  Change at DC Week 1 (n=109,30,94,29,99,30) | -11.0 (9.48) | -12.9 (7.89) | -11.0 (8.08) | -9.9 (10.98) | -8.7 (10.77) | -10.4 (7.58)
  Change at DC Week 2 (n=106,29,84,26,92,30) | -9.8 (10.32) | -13.8 (8.32) | -10.8 (8.42) | -10.2 (8.56) | -9.6 (9.70) | -10.3 (7.50)

22. Secondary Outcome: Physician's Withdrawal Checklist (PWC) Score for Cohort 1 (Less Than 3-Month Last Visit)
Description: as for outcome 7
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 19 | 18
units on a scale
  Discontinuation Week 1 (n=15,19,18) | 10.2 (7.97) | 14.3 (10.04) | 9.1 (9.25)
  Discontinuation Week 2 (n=14,15,16) | 8.2 (6.70) | 14.1 (9.16) | 10.6 (9.39)

23. Secondary Outcome: Physician's Withdrawal Checklist (PWC) Score for Cohort 2 (3-Month Last Visit)
Description: as for outcome 7
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 49
units on a scale
  Discontinuation Week 1 (n=58,52,49) | 9.1 (6.82) | 8.0 (6.19) | 7.3 (6.69)
  Discontinuation Week 2 (n=54,49,44) | 8.9 (7.28) | 8.3 (6.32) | 6.9 (6.38)

24. Secondary Outcome: Physician's Withdrawal Checklist (PWC) Score for Cohort 3 (6-Month Last Visit)
Description: as for outcome 7
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included. N (Number of Participants Analyzed) = participants evaluable for this measure. 'n' = participants evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 29 | 99 | 30
units on a scale
  Discontinuation Week 1 (n=109,30,94,29,99,30) | 6.8 (6.56) | 4.9 (5.73) | 5.1 (4.45) | 7.4 (6.43) | 8.0 (7.45) | 4.6 (4.22)
  Discontinuation Week 2 (n=106,29,84,26,93,30) | 7.9 (7.59) | 4.1 (4.17) | 5.7 (6.11) | 7.1 (8.65) | 7.1 (6.64) | 4.6 (4.67)

25. Secondary Outcome: Change From Last Visit of Treatment in Hamilton Anxiety Scale (HAM-A) for Cohort 1 (Less Than 3-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 1
Time Frame: Last visit on treatment, Week 1, 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 18 | 20
units on a scale
  Last visit on treatment (n=15,18,20) | 16.1 (8.46) | 21.6 (6.18) | 16.1 (10.11)
  Change at Discontinuation Week 1 (n=15,18,18) | 2.0 (11.45) | -2.3 (4.63) | -2.4 (3.31)
  Change at Discontinuation Week 2 (n=14,15,16) | -2.3 (9.47) | -3.5 (5.34) | -2.2 (4.18)

26. Secondary Outcome: Change From Last Visit of Treatment in Hamilton Anxiety Scale (HAM-A) for Cohort 2 (3-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 6
Time Frame: Last visit on treatment, Week 1, 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 50
units on a scale
  Last visit on treatment (n=58,52,50) | 8.0 (6.57) | 8.5 (6.50) | 6.7 (4.29)
  Change at Discontinuation Week 1 (n=58,52,48) | 1.7 (6.69) | 0.9 (4.03) | 2.3 (5.74)
  Change at Discontinuation Week 2 (n=54,49,44) | 1.5 (5.55) | 1.5 (6.43) | 1.5 (5.37)

27. Secondary Outcome: Change From Last Visit of Treatment in Hamilton Anxiety Scale (HAM-A) for Cohort 3 (6-Month Last Visit) at Discontinuation Week 1 and 2
Description: as for outcome 1
Time Frame: Last visit on treatment, Week 1, 2 post-treatment discontinuation (discontinuation [DC] occurred after Week 15 to Week 24)
Population: Per-protocol analysis set. Cohort 3: Participants who discontinued study after Week 15 or completed Week 24 visit and had at least 1 discontinuation assessment were included. N(Number of Participants Analyzed) = participants evaluable for this measure. 'n' = participants evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 93 | 29 | 100 | 30
units on a scale
  Last visit on treatment (n=109,30,93,29,100,30) | 6.3 (5.89) | 5.5 (6.12) | 5.6 (5.02) | 8.3 (6.49) | 5.6 (6.17) | 5.5 (4.66)
  Change at DC Week 1 (n=109,30,93,28,99,30) | 1.6 (4.37) | -0.0 (2.30) | 0.7 (3.08) | 0.6 (2.69) | 3.0 (5.73) | 0.3 (3.01)
  Change at DC Week 2 (n=107,29,84,26,94,30) | 2.5 (5.74) | -0.8 (5.33) | 1.2 (3.90) | 1.5 (5.08) | 2.2 (5.39) | 0.6 (3.76)

28. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) for Cohort 1 (Less Than 3-Month Last Visit)
Description: as for outcome 1
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation occurred prior to Week 9)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 15 | 19 | 18
units on a scale
  Discontinuation Week 1 (n=15,19,18) | 18.1 (7.11) | 19.0 (7.61) | 14.1 (10.31)
  Discontinuation Week 2 (n=14,15,16) | 13.9 (7.33) | 18.6 (6.15) | 14.6 (10.41)

29. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) for Cohort 2 (3-Month Last Visit)
Description: as for outcome 6
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation occurred from Week 9 to Week 15)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 58 | 52 | 48
units on a scale
  Discontinuation Week 1 (n=58,52,48) | 9.6 (6.38) | 9.4 (6.60) | 8.8 (5.88)
  Discontinuation Week 2 (n=54,49,44) | 9.0 (6.44) | 9.9 (7.04) | 8.3 (6.48)

30. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) Score for Cohort 3 (6-Month Last Visit)
Description: as for outcome 1
Time Frame: Week 1, 2 post-treatment discontinuation (discontinuation [DC] occurred after Week 15 to Week 24)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 109 | 30 | 94 | 28 | 99 | 30
units on a scale
  Discontinuation Week 1 (n=109,30,94,28,99,30) | 7.9 (6.34) | 5.5 (4.85) | 6.3 (5.48) | 8.4 (6.67) | 8.4 (7.07) | 7.07 (4.92)
  Discontinuation Week 2 (n=107,29,84,26,94,30) | 8.9 (7.60) | 5.0 (4.32) | 6.5 (6.36) | 9.2 (8.28) | 7.9 (6.27) | 6.1 (6.00)

31. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) Score for Period 1
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 197 | 183 | 188
units on a scale
  Baseline | 25.3 (4.39) | 24.9 (3.87) | 24.5 (4.39)
  Week 12 | 8.0 (6.23) | 8.9 (7.19) | 7.9 (6.70)

32. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) Score for Period 2
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 117 | 37 | 103 | 37 | 106 | 37
units on a scale
  Baseline | 25.6 (3.82) | 24.6 (4.66) | 24.8 (3.77) | 25.1 (3.92) | 24.7 (4.41) | 24.1 (4.03)
  Week 24 | 7.0 (6.53) | 7.1 (7.09) | 6.5 (5.98) | 10.2 (7.49) | 5.7 (6.06) | 6.6 (6.33)

33. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Score at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. LOCF method was used to impute missing values. Here, N (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 194 | 180 | 185
units on a scale | -17.4 (7.39) | -16.0 (7.45) | -16.7 (7.92)

34. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Score at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 117 | 37 | 103 | 37 | 106 | 37
units on a scale | -18.7 (7.33) | -17.5 (6.89) | -18.2 (6.59) | -14.9 (7.85) | -19.0 (7.24) | -17.5 (8.34)

35. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score for Period 1
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 197 | 183 | 188
units on a scale
  Baseline | 4.6 (0.68) | 4.5 (0.71) | 4.4 (0.65)
  Week 12 | 2.3 (1.06) | 2.5 (1.17) | 2.3 (1.00)

36. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score for Period 2
Description: as for outcome 35
Time Frame: Baseline, Week 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 117 | 37 | 103 | 37 | 106 | 37
units on a scale
  Baseline | 4.7 (0.65) | 4.5 (0.69) | 4.5 (0.71) | 4.5 (0.73) | 4.4 (0.68) | 4.5 (0.56)
  Week 24 | 2.3 (1.08) | 2.2 (1.16) | 2.1 (0.97) | 2.5 (1.24) | 1.9 (0.90) | 2.4 (0.98)

37. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 12
Description: as for outcome 35
Time Frame: Baseline, Week 12
Population: Per-protocol analysis set: all randomized participants who had baseline with at least 1 discontinuation or efficacy visit, and were not major protocol violators. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 195 | 181 | 186
units on a scale | -2.3 (1.13) | -2.1 (1.13) | -2.1 (1.17)

38. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 24
Description: as for outcome 35
Time Frame: Baseline, Week 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 117 | 37 | 103 | 37 | 106 | 37
units on a scale | -2.4 (1.13) | -2.3 (1.24) | -2.4 (1.04) | -2.0 (1.27) | -2.5 (1.11) | -2.2 (1.17)

39. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score at the End of Period 1
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale.
Time Frame: Week 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 197 | 183 | 188
units on a scale | 1.9 (1.13) | 1.9 (1.01) | 1.9 (1.17)

40. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score at the End of Period 2
Description: as for outcome 39
Time Frame: Week 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 117 | 37 | 103 | 37 | 106 | 37
units on a scale | 1.7 (0.99) | 1.9 (1.15) | 1.6 (0.75) | 2.3 (1.53) | 1.5 (0.91) | 2.0 (1.07)

41. Other Pre Specified Outcome: Sheehan-Suicidality Tracking Scale (S-STS) Score
Description: Sheehan-Suicidality Tracking Scale (S-STS): an 8-item prospective rating scale that tracked treatment-emergent suicidal ideation and behaviors. Items 1a, 2-6, 7a, and 8 were scored on a 5-point Likert scale (ranging from 0= not at all to 4=extremely). Items 1, 1b, and 7 required yes or no responses. Total score ranged from 0 to 35, higher score indicated higher suicidal tendency.
Time Frame: Baseline up to Week 24
Population: Data was not statistically summarized but was available in individual participant listings and mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) due to change in planned analysis.
Arm/Group | Pregabalin High Dose | Pregabalin Low Dose | Lorazepam
Number analyzed (Participants) | 0 | 0 | 0

42. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and Week 12, for period 1, and between Week 13 and Week 24, for period 2, that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Week 12 (period 1), Week 13 up to Week 24 (period 2)
Population: Safety analysis set: all randomized participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable for this measure during each specified period, for each group respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Number analyzed (Participants) | 154 | 52 | 154 | 52 | 153 | 50
participants
  Period 1 (n=154,52,154,52,153,50) | 103 | 37 | 100 | 40 | 95 | 35
  Period 2 (n=121,39,112,38,114,39) | 62 | 26 | 62 | 18 | 52 | 20

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin High Dose, Pregabalin High Dose | Pregabalin High Dose, Placebo | Pregabalin Low Dose, Pregabalin Low Dose | Pregabalin Low Dose, Placebo | Lorazepam, Lorazepam | Lorazepam, Placebo
Serious Adverse Events (participants affected / at risk) | 2/154 | 0/52 | 5/154 | 2/52 | 4/153 | 0/50
Other Adverse Events (participants affected / at risk) | 110/154 | 40/52 | 108/154 | 38/52 | 100/153 | 35/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin High Dose, Pregabalin High Dose (N=154) | Pregabalin High Dose, Placebo (N=52) | Pregabalin Low Dose, Pregabalin Low Dose (N=154) | Pregabalin Low Dose, Placebo (N=52) | Lorazepam, Lorazepam (N=153) | Lorazepam, Placebo (N=50)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin High Dose, Pregabalin High Dose (N=154) | Pregabalin High Dose, Placebo (N=52) | Pregabalin Low Dose, Pregabalin Low Dose (N=154) | Pregabalin Low Dose, Placebo (N=52) | Lorazepam, Lorazepam (N=153) | Lorazepam, Placebo (N=50)
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 5 | 4 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 10 | 1 | 4 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | 8 | 5 | 9 | 1
Dry mouth (Gastrointestinal disorders) | 13 | 3 | 5 | 2 | 8 | 4
Nausea (Gastrointestinal disorders) | 17 | 7 | 12 | 8 | 18 | 7
Fatigue (General disorders) | 16 | 6 | 15 | 11 | 15 | 5
Irritability (General disorders) | 6 | 1 | 4 | 2 | 8 | 1
Influenza (Infections and infestations) | 8 | 3 | 7 | 0 | 7 | 0
Nasopharyngitis (Infections and infestations) | 13 | 2 | 7 | 5 | 8 | 4
Weight increased (Investigations) | 5 | 1 | 7 | 3 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 3 | 4 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 1 | 0 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 2 | 9 | 1
Disturbance in attention (Nervous system disorders) | 12 | 1 | 3 | 2 | 6 | 1
Dizziness (Nervous system disorders) | 37 | 17 | 28 | 14 | 20 | 10
Headache (Nervous system disorders) | 38 | 13 | 36 | 17 | 33 | 10
Paraesthesia (Nervous system disorders) | 6 | 0 | 3 | 3 | 5 | 2
Sedation (Nervous system disorders) | 6 | 2 | 5 | 0 | 10 | 1
Somnolence (Nervous system disorders) | 25 | 7 | 31 | 9 | 35 | 13
Tremor (Nervous system disorders) | 5 | 2 | 1 | 3 | 6 | 0
Anxiety (Psychiatric disorders) | 14 | 6 | 10 | 1 | 19 | 5
Generalised anxiety disorder (Psychiatric disorders) | 4 | 2 | 9 | 2 | 6 | 2
Insomnia (Psychiatric disorders) | 31 | 15 | 24 | 12 | 23 | 13
Tension (Psychiatric disorders) | 8 | 1 | 4 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.